CLINICAL TRIAL: NCT02799719
Title: Body Fat Mass as Predictors of Survival in Hemodialysis Patients and Its Association With Clinical Metabolic Profiles, Markers of Inflammation and Adipocytokines in Chronic Hemodialysis Patients: a Prospective Study.
Brief Title: Body Fat Mass Association With Clinical Metabolic Profiles, Markers of Inflammation and Adipocytokines
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102047
Record Dates: First submitted 2016-05-26; First posted 2016-06-15 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Overweight and Obesity
Keywords: Fat mass; hemodialysis patients; inflammation; adipocytokines; bioimpedance spectroscopy
MeSH Terms: conditions — Overweight; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Overweight and obesity have become an increasing problem in patients on hemodialysis. However, in virtually all observational studies in chronic kidney disease(CKD) and dialysis patients , using body mass index(BMI) as metric fat mass is associated inversely with death rate. Nevertheless, it is questionable that obesity can be considered an unequivocal protective factor in chronic diseases as increase body fat mass appears to be a potential cause of the chronic inflammation frequently present in these patients. The consequences of this inflammation are impaired nutritional status, accelerated atherosclerosis, and increased mortality. In the present study, by using dual-energy X-ray absorptiometry (DEXA) and bioimpedance spectroscopy (BIS) to evaluated the contributions of fat mass to outcomes in an observational cohort of hemodialysis patients. Besides, we aim to assess the relationship between body fat composition, clinical metabolic risk profiles, measures of adiposity, such as waist circumference (WC), visceral adiposity index, waist-to-hip ratio (WHR), and waist-to-height ratio (WHtR), markers of inflammation and adipocytokines in these maintenance hemodialysis patients.

DETAILED DESCRIPTION:
Patient Selection

Clinically stable stage 5 chronic kidney disease patients (400 patients) attending the Tungs Taichung Metroharbour will be enrolled in this study. These patients will be given written information and are invited to participate in the study. Written informed consent will be obtained from each patient enrolled. Our hospital dialysis center undergoes multi-frequency bioelectrical impedance analysis( BIA) scanning on a bimonthly basis as part of their ongoing clinical care. Multi-frequency BIA is performed on patients attending the center as part of their routine dry weight assessment. Among these patients, eighty ambulatory adults attending for thrice-weekly outpatient hemodialysis treatments concomitantly had similar dual-energy X-ray absorptiometry (DEXA) scan and postdialysis multi-frequency BIA assessments for review. Patients with implantable defibrillators, those with cardiac pacemakers, and amputees are excluded from the study. This study will be conducted prospectively for 3 years.

Methods Body Composition Assessment Measurements with dual-energy X-ray absorptiometry (DEXA)

DEXA was performed with patients in the supine position. The radiation exposure is estimated to be one tenth of that for standard chest radiography. DEXA is scheduled postdialysis. Whole-body composition, including total and segmental lean, total body fat mass, and bone mineral content, will be calculated using the compatible software. For patients with multiple multifrequency BIA estimations, the study performed will be arranged temporally to the DEXA scan for more relevant comparison.

Measurement of Bioimpedance In all patients BIS will be carried out bimonthly using the Body Composition Monitor (Fresenius Medical Care Deutschland Gesellschaft mit beschrankter Haftung (GmbH), Germany), which takes measurements at 50 frequencies in a range of 5 to 1000 kilohertz(KHz). The measurement was performed approximately 30 minutes after the midweek hemodialysis session, with four conventional electrodes being placed in the patient, who was lying in the supine position: two in the hand and two in the foot contralateral to the vascular access. Regarding the quality of measurements, all exceeded 95%. The manufacturer of the Body Composition Monitor (Fresenius Medical Care) indicated that 30 minutes after the hemodialysis session, the balance between intra-and extracellular fluid was restored and no significant differences in relation to pre-dialysis values were observed. Parameters obtain directly through BIS that are used in this study are free fat mass, lean body mass, intracellular water (ICW) and extracellular water( ECW). Protein-energy wasting (PEW), represented by the intracellular water/dry body weight (ICW/BW) ratio, and overhydration, represented by the extracellular water/dry body weight(ECW/BW) ratio will be analysed.

Anthropometric parameters The following data will collected bimonthly : height (m)), dry weight (kg) measured with a calibrated scale and body mass index(BMI,kg/m2). Abdominal obesity is defined as a waist circumference of >80 cm in women and >90 cm in men.

Biochemical assays and other measurements Fasting blood samples (4 ml each time) were taken just before starting a dialysis session.The vacutainers were kept cold and placed immediately on ice, then they were centrifuged at 4 degree centigrade and the serum was stored at -80 degree centigrade until the analysis. The measurements of serum creatinine, cholesterol, total proteins, albumin, prealbumin and carbon dioxide(CO2) were analysed using standard methods. Urea reduction ratio and single-pool dialysis efficiency calculator(Kt/V) were used to represent the administered dialysis treatment dose. To decrease intraindividual variation, 3-month averaged values for laboratory measures and urea reduction ratio during the study calendar quarter were calculated and used in this study. High sensitivity C- reactive proteins(CRP) was obtained by the immuno-turbidimetric method. Serum 25(OH)D3 was measured by enzymeimmunoassay and the levels of intact parathyroid hormone( i-PTH) were assessed using immunoradiometric assay. Plasma insulin levels were measured using a radioimmunoassay method. Interleukin-6(IL-6) and tumor necrosis factor-alpha (TNF-α) concentrations were measured in duplicate by enzyme-linked immunosorbent assay(ELISA). Insulin resistance was assessed using the following validated formula: homeostasis model assessment of insulin resistance (HOMA-IR)=(fasting glucose [mmol/1] × fasting insulin [μU/ml])/22.5. Because of confounding introduced by exogenous insulin administration to HOMA-IR results, HOMA-IR was only measured in patients who were not treated with insulin . All the above measurements will be done at baseline, and the end of each years (4 times for the whole study)

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged > 20 years-old. Received stable hemodialysis at least 3 months. Written informed consent.

Exclusion Criteria:

* Patients with malignant disease, acute infectious disease, acute inflammatory disease (such as collagen disease), and advanced liver disease are excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Occurence of CVD events | 3 years
  A DEXA scan is used to measure total and segmental lean(kg), total body fat mass(kg), and bone mineral content(kg).
  A BIS is used to measurefree fat mass(Kg), lean body mass(Kg),ICW(L) and ECW(L).

SECONDARY OUTCOMES:
Correlates of metabolic syndrome | 3 years
  The measurements of cholesterol(mg/dl),albumin(mg/dl) ,plasma insulin levels(mU/L) were measured using a radioimmunoassay method. Insulin resistance was assessed using the following validated formula: homeostasis model assessment of insulin resistance (HOMA-IR)=(fasting glucose [mmol/1] × fasting insulin [μU/ml])/22.5
Presence of inflammation | 3 years
  Various biomarkers such as CRP, IL-6, TNF-a

IPD SHARING:
Plan to Share IPD: Yes